CLINICAL TRIAL: NCT07312552
Title: The Impact of Periodontal Status and Smoking on Salivary Inflammasome Levels: A Cross-Sectional Study
Brief Title: Association of Periodontal Status and Smoking With Salivary Inflammasome Markers
Status: Recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Kubra Karaduran, Assistant Professor, Uskudar University
Other Study IDs: KKARADURAN1
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis; Periodontal Disease; Periodontal Health; Smoking; Inflammasomes
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Unstimulated whole saliva samples will be collected from all participants. Samples will be stored at -80°C until analysis.The stored saliva samples will be used exclusively for the measurement of biomarker levels via ELISA. No DNA extraction or genetic analyses will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 (C): Healthy individuals (control (C))
  Interventions: Diagnostic Test: Periodontal examinations; Diagnostic Test: Collection of saliva samples
- Group 2 (S-C): Smokers with healthy periodontium (S-C)
  Interventions: Diagnostic Test: Periodontal examinations; Diagnostic Test: Collection of saliva samples
- Group 3 (P): Nonsmokers with Stage III/IV periodontitis (P)
  Interventions: Diagnostic Test: Periodontal examinations; Diagnostic Test: Collection of saliva samples
- Group 4 (S-P): Smokers with Stage III/IV periodontitis (S-P)
  Interventions: Diagnostic Test: Periodontal examinations; Diagnostic Test: Collection of saliva samples

INTERVENTIONS:
Diagnostic Test: Periodontal examinations — With periodontal evaluation, plaque percentage, probing pocket depth, percentage of bleeding on probing, clinical attachment level, number of teeth, periodontal inflammatory surface area (PISA) parameters are recorded.
Diagnostic Test: Collection of saliva samples — Levels of salivary NOD-like receptor family, pyrin domain containing 3 (NLRP-3), NOD-like receptor family, pyrin domain containing 6 (NLRP-6), NOD-like receptor family, pyrin domain containing 12 (NLRP-12), NOD-like receptor family, CARD domain containing 5 (NLRC-5), interleukin-1 beta (IL-1β), and interleukin-10 (IL-10) will be determined using an enzyme-linked immunosorbent assay (ELISA).

SUMMARY:
The aim of this study is to evaluate the relationship between periodontal status and salivary levels of the inflammasomes NOD-like receptor family, pyrin domain containing 3 (NLRP-3), NOD-like receptor family, pyrin domain containing 6 (NLRP-6), NOD-like receptor family, pyrin domain containing 12 (NLRP-12), NOD-like receptor family, CARD domain containing 5 (NLRC-5), interleukin-1 beta (IL-1β) and interleukin-10 (IL-10). Furthermore, this study aims to investigate whether the salivary levels of these inflammasomes may serve as potential diagnostic biomarkers for distinguishing individuals with periodontitis from those without. In addition, the potential role of smoking in modulating the relationship between periodontal status and salivary inflammasome levels will also be explored.

DETAILED DESCRIPTION:
The aim of this study was to determine the periodontal status and smoking status of the participants, to obtain clinical periodontal records and to explain their relationship with salivary NLRP-3 NLRP-6, NLRP-12, NLRC-5, IL-1β and IL-10 levels.

The participants included in the study will be divided into four groups: smokers with periodontal disease, non-smokers with periodontal disease, smokers without periodontal disease, and non-smokers without periodontal disease. Systemic and dental anamnesis of the participants will be taken, smoking habits will be evaluated, medical records and current diagnoses will be examined, intraoral examinations will be performed and periodontal records will be taken. The periodontal status of the participants will be diagnosed according to the 'Classification of Periodontal and Peri-implant Diseases and Conditions' accepted at the 2017 World Workshop, supported by the American Academy of Periodontology (AAP) and the European Federation of Periodontology (EFP).

Saliva samples will be collected before clinical periodontal measurements. The collected saliva samples will be stored at -80°C until analyzed. Salivary NLRP-3, NLRP-6, NLRP-12, NLRC-5, IL1β, and IL-10 levels will be measured using an enzyme-linked immunosorbent assay (ELISA) method.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy,
* clinical diagnosis of periodontitis,
* clinical diagnosis of periodontal health

Exclusion Criteria:

* history of regular use of systemic antibiotics, anti-inflammatory, or antioxidant drugs (previous 6 months);
* nonsurgical periodontal treatment (previous 6 months);
* surgical periodontal treatment (previous 12 months);
* presence of <20 teeth;
* current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy);
* diabetes diagnosis; rheumatoid arthritis diagnosis; and pregnancy, lactating, or excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will consist of four groups:
  Group 1: healthy individuals (control (C)), Group 2: smokers with healthy periodontium (S-C), Group 3: nonsmokers with Stage III/IV periodontitis (P), Group 4: smokers with Stage III/IV periodontitis (S-P)
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (mm) | Baseline
  Clinical attachment level (CAL) is a more reliable indicator of periodontal support around a tooth than probing depth alone, as it is measured from a fixed anatomical landmark-the cementoenamel junction (CEJ)-which remains constant over time.
  Calculating CAL requires two measurements: the distance from the gingival margin to the CEJ and the probing depth.
  In cases of gingival recession, CAL is calculated by adding the probing depth to the distance from the gingival margin to the CEJ.
  In cases of gingival overgrowth, CAL is determined by subtracting the distance from the gingival margin to the CEJ from the probing depth.
Probing pocket depth | Baseline
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Bleeding on probing | Baseline
  The number obtained by dividing the sum of the positive areas by the sum of the examined areas is multiplied by 100 and the value obtained is expressed as the percentage of bleeding at probing (BOP%).

SECONDARY OUTCOMES:
Plaque percentage | Baseline
  The presence or absence of plaque is determinant, recorded as (+) in the presence of plaque or (-) in the absence of plaque, and the percentage of the entire mouth affected by plaque is expressed as a percentage (P%).
Periodontal inflammatory surface area (PISA) | Baseline
  It is the calculation of the area of ulcerated periodontal pockets showing bleeding on probing based on the periodontal epithelial surface area.
Salivary interleukin-10 (IL-10) levels | Baseline
  Saliva samples will be collected prior to clinical periodontal measurements. The collected saliva samples will be stored at -80°C until analysis. Il-10 levels in saliva will be measured using the enzyme-linked immunosorbent assay (ELISA) method.
Salivary interleukin-1beta (IL-1β) levels | Baseline
  Saliva samples will be collected prior to clinical periodontal measurements. The collected saliva samples will be stored at -80°C until analysis. IL-1β levels in saliva will be measured using the ELISA method.
Salivary NOD-like receptor family, pyrin domain containing 3 (NLRP-3) levels | Baseline
  Saliva samples will be collected prior to clinical periodontal measurements. The collected saliva samples will be stored at -80°C until analysis. NLRP-3 levels in saliva will be measured using the ELISA method.
Salivary NOD-like receptor family, pyrin domain containing 6 (NLRP-6) levels | Baseline
  Saliva samples will be collected prior to clinical periodontal measurements. The collected saliva samples will be stored at -80°C until analysis. NLRP-6 levels in saliva will be measured using the ELISA method.
Salivary NOD-like receptor family, pyrin domain containing 12 (NLRP-12) levels | Baseline
  Saliva samples will be collected prior to clinical periodontal measurements. The collected saliva samples will be stored at -80°C until analysis. NLRP-12 levels in saliva will be measured using the ELISA method.
Salivary NOD-like receptor family, CARD domain containing 5 (NLRC-5) levels | Baseline
  Saliva samples will be collected prior to clinical periodontal measurements. The collected saliva samples will be stored at -80°C until analysis. NLRC-5 levels in saliva will be measured using the ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra KARADURAN, Principal Investigator — Uskudar University
Locations (1):
- Uskudar University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)